CLINICAL TRIAL: NCT00415207
Title: Pharmacogenomics of Paclitaxel in Ovarian Cancer: Predictors of Toxicity and Response
Brief Title: Pharmacogenomics of Paclitaxel in Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Danish Clinical Intervention Research Academy (Other); Ministry of the Interior and Health, Denmark (Other Government)
Responsible Party: Troels K Bergmann, University of Southern Denmark
Other Study IDs: WRAMC WU# 04-23009
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2006-12

CONDITIONS: Ovarian Neoplasms; Fallopian Tube Neoplasms
Keywords: CYP2C8; MDR1; Pharmacogenetics; Paclitaxel
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — paraffin embedded biopsies

SUMMARY:
This study will try to determine whether or not certain genes are responsible for the huge variation in toxicity and effect observed between patients treated with paclitaxel (chemotherapeutic drug). Specifically we will study this retrospectively in patients who participated in clinical trials that are now closed. All patients had ovarian cancer and received paclitaxel/carboplatin chemotherapy after primary surgery.

DETAILED DESCRIPTION:
Paclitaxel is an antineoplastic drug used in the treatment of ovarian cancer. The effect and toxicity is unpredictable in the individual patient. Paclitaxel is removed (eliminated) from the organism by oxidation. CYP2C8 is the enzyme mainly responsible. P-glycoprotein (Pgp) is an efflux transport protein natural to the human organism. Pgp is responsible for excretion of drugs via the bile and the kidneys and is thought to play a role in chemotherapy resistance. Paclitaxel is substrate for Pgp. Single nucleotide polymorphisms are possible causes for variation in both CYP2C8 and Pgp expression/function. We will study a possible role of these genetic variations as predictors of paclitaxel toxicity and effect and the possible implications for individual dosing in the future.

We will use tissue from patients who participated in one of two clinical trials that are both closed for inclusion. Genotypic data from this tissue will be correlated with toxicity and survival data drawn from a research database. We expect to be able to find >300 available cases to study.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in "TC/TEC" in Denmark, Sweden or Norway
* Patients enrolled in "OVAR-9" in Denmark, Sweden or Norway

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2006-12; Primary Completion 2008-08 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Brøsen, phd, Study Director — University of Southern Denmark
Locations (1):
- Clinical Pharmacology, University of Southern Denmark, Odense, Denmark

REFERENCES:
- [Result] Bergmann TK, Green H, Brasch-Andersen C, Mirza MR, Herrstedt J, Holund B, du Bois A, Damkier P, Vach W, Brosen K, Peterson C. Retrospective study of the impact of pharmacogenetic variants on paclitaxel toxicity and survival in patients with ovarian cancer. Eur J Clin Pharmacol. 2011 Jul;67(7):693-700. doi: 10.1007/s00228-011-1007-6. Epub 2011 Feb 16. PMID 21327421